CLINICAL TRIAL: NCT04610164
Title: The Effect of Tranexamic Acid on Visualization During Shoulder Arthroscopy
Brief Title: The Effect of Tranexamic Acid (TXA) on Visualization During Shoulder Arthroscopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNAM18d.610
Record Dates: First submitted 2020-10-21; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Shoulder Arthroscopy; Operative Bleeding; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: TXA group (Experimental): Patient will receive 1 gram intravenous TXA prior to surgery
  Interventions: Drug: Tranexamic acid
- Group 2: Control Group (No Intervention): Patient will not receive TXA prior to surgery

INTERVENTIONS:
Drug: Tranexamic acid — Prior to surgery, the patient will receive 1 gram of IV TXA
  Arms: Group 1: TXA group

SUMMARY:
Tranexamic acid has seen an increase in use over the past decade in hip and knee arthroplasty as well as spine surgery with more recent use seen in total shoulder arthroplasty (TSA). The mechanism of action of TXA is as a lysine analogue that competitively inhibits the conversion of plasminogen to plasmin thus resulting in its antifibrinolytic activity. Investigators have showed that compared with placebo TXA had a statistically significant effect on blood and postoperative hemoglobin levels in TSA. To date there are no studies investigating the effect of TXA in arthroscopy of any kind or studies examining the ability of TXA to aid in surgeon visualization in arthroscopic procedures. The investigators of this study will use change in pump pressure as a surrogate objective measure for surgeon visualization. The hypothesis is that participants who receive TXA will have a lower change in pump pressure compared to participants who do not receive TXA.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 18-80
* participants with an ASA (American Society of Anesthesiologists) score 1-3
* participants with a surgical indication of full thickness small to massive rotator cuff tear.

Exclusion Criteria:

* pregnant females,
* participants with a known allergy to tranexamic acid,
* participants with active thromboembolic disease,
* participants with seizure disorder,
* participants with prior cerebrovascular accident (CVA),
* history of cardiac stents or past history of thromboembolic disease,
* presence of full-thickness subscapularis tear (>50%),
* participants with irreparable rotator cuff tears.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in operative factors | 2 hours
  change in pump pressure (ΔP) during shoulder arthroscopy with a change in pump pressure of 15 mmHg set as the marker of surgeon visualization of the shoulder joint during surgery.
Postoperative pain | 7 days
  Investigators will be measuring whether there is a decrease in participants pain after surgery as assessed by visual analog score 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States